CLINICAL TRIAL: NCT01276457
Title: An 18 Month Extension to the Multicenter, Randomized, Open-label Trial (NCT00170885) to Evaluate the Safety, Tolerability, and Efficacy of Two Regimens of Everolimus Plus Cyclosporine Microemulsion, Given According to Different Blood Target Levels, in de Novo Renal Transplant Recipients
Brief Title: Everolimus in Combination With Cyclosporine Microemulsion in de Novo Renal Transplant Recipients
Acronym: EVEREST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001AIT02E1
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Results first posted 2011-04-19 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-05

CONDITIONS: Transplantation Infection
Keywords: immunosuppression; kidney transplantation; everolimus; safety
MeSH Terms: interventions — Cyclosporine

ARMS (2):
- Upper everolimus blood target + very low dose cyclosporine (Experimental): Patients received everolimus orally twice daily at a dose that was adjusted to achieve a drug blood trough level in the range of 8-12 ng/mL. Patients also received a very low dose of cyclosporine (150-300 ng/mL) orally twice daily that was adjusted to maintain a drug blood level of 200 ng/mL 2 hours after the morning dose. Both drugs were taken in the morning and again 12 hours later. The drugs were taken consistently either before, during, or after meals. No grapefruit or grapefruit juice was allowed throughout the study.
  Interventions: Drug: Everolimus 0.25 and 0.75 mg tablets; Drug: Cyclosporine very low dose (150-300 ng/mL) microemulsion
- Standard everolimus blood target + low dose cyclosporine (Active Comparator): Patients received everolimus orally twice daily at a dose that was adjusted to achieve a drug blood trough level in the range of 3-8 ng/mL. Patients also received a low dose of cyclosporine (350-500 ng/mL) orally twice daily that was adjusted to maintain a drug blood level of 400 ng/mL 2 hours after the morning dose. Both drugs were taken in the morning and again 12 hours later. The drugs were taken consistently either before, during, or after meals. No grapefruit or grapefruit juice was allowed throughout the study.
  Interventions: Drug: Everolimus 0.25 and 0.75 mg tablets; Drug: Cyclosporine low dose (350-500 ng/mL) microemulsion

INTERVENTIONS:
Drug: Everolimus 0.25 and 0.75 mg tablets — The dose of everolimus for each patient was adjusted to achieve the target everolimus blood level range. Everolimus blood trough level was measured 5 days after any dose adjustment to verify that the blood level was within the desired target level range.
Drug: Cyclosporine very low dose (150-300 ng/mL) microemulsion — The dose of cyclosporine for each patient was adjusted to achieve the target cyclosporine blood level. Cyclosporine dose adjustments were based on drug blood level determined from whole blood samples taken 2 hours (± 10 min) after the morning dose.
  Other Names: Neoral
  Arms: Upper everolimus blood target + very low dose cyclosporine
Drug: Cyclosporine low dose (350-500 ng/mL) microemulsion — The dose of cyclosporine for each patient was adjusted to achieve the target cyclosporine blood level. Cyclosporine dose adjustments were based on drug blood level determined from whole blood samples taken 2 hours (± 10 min) after the morning dose.
  Other Names: Neoral
  Arms: Standard everolimus blood target + low dose cyclosporine

SUMMARY:
The purpose of this study was to allow the continuation of everolimus treatment in patients who have completed the core study (NCT00170885) and to collect long-term safety, tolerability, and efficacy data in a group of patients treated with the upper everolimus target levels plus very low dose cyclosporin in comparison with the standard everolimus target levels plus low dose cyclosporin in patients with renal transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with functioning graft who had completed the 6-month treatment period of core study
* Patients who were receiving treatment with either everolimus and cyclosporin at the end of the core study
* Patients who signed the informed consent of the present study extension

Exclusion Criteria:

- Women who were pregnant, lactating or who wished to became pregnant.

Other protocol-defined inclusion/exclusion criteria applied to the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2006-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was an 18-month extension to the 6-month core study NCT01276457. All patients who were receiving treatment at the end of the core study and signed the informed consent of the extension study were included. Patients received the same treatment in the extension study that they received in the core study.
Period: Core Study
Arm/Group | Upper Everolimus Blood Target + Very Low Dose Cyclosporine | Standard Everolimus Blood Target + Low Dose Cyclosporine
Started | 142 | 143
Completed | 129 | 123
Not Completed | 13 | 20
Not completed — Adverse Event | 6 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Administrative problems | 1 | 1
Not completed — Death | 2 | 2
Not completed — Lack of Efficacy | 3 | 12
Period: Extension Study
Arm/Group | Upper Everolimus Blood Target + Very Low Dose Cyclosporine | Standard Everolimus Blood Target + Low Dose Cyclosporine
Started | 111 | 112
Completed | 105 | 110
Not Completed | 6 | 2
Not completed — Lost to Follow-up | 3 | 0
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Upper Everolimus Blood Target + Very Low Dose Cyclosporine | Standard Everolimus Blood Target + Low Dose Cyclosporine | Total
Number analyzed (Participants) | 111 | 112 | 223
Age Continuous [Mean (Standard Deviation); unit: Years] | 45.3 (12.2) | 45.7 (10.2) | 45.5 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 37 | 77
  Male | 71 | 75 | 146

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Biopsy-proven Acute Rejection
Description: A graft core biopsy was performed on all suspected acute rejection episodes within 48 hours. Biopsies were read by the local pathologist according to the 1997 Banff criteria. A biopsy-proven acute rejection was be defined as a biopsy graded IA, IB, IIA, IIB, or III.
Time Frame: Baseline to end of study (Month 24)
Population: Intent-to-treat (ITT) population: All randomized subjects for whom at least one valid post-baseline efficacy measurement was obtained and used for efficacy analyses.
Measure: Number; unit: Participants
Arm/Group | Upper Everolimus Blood Target + Very Low Dose Cyclosporine | Standard Everolimus Blood Target + Low Dose Cyclosporine
Number analyzed (Participants) | 142 | 143
Participants | 21 | 21

2. Primary Outcome: Renal Function Assessed by Creatinine Clearance
Description: Renal function was assessed by measuring serum creatinine and by computing creatinine clearance using the formula of Cockcroft-Gault.
Time Frame: Month 12, Month 18, and Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Upper Everolimus Blood Target + Very Low Dose Cyclosporine | Standard Everolimus Blood Target + Low Dose Cyclosporine
Number analyzed (Participants) | 111 | 111
mL/min
  Month 12 (n=111, 111) | 61.26 (22.06) | 62.50 (20.70)
  Month 18 (n=108, 108) | 60.90 (22.85) | 62.80 (21.18)
  Month 24 (n=106, 110) | 61.92 (25.37) | 63.76 (21.71)

3. Secondary Outcome: Number of Participants Who Died, Number of Participants Who Lost Their Graft, and Number of Participants Who Died or Lost Their Graft
Description: A participant lost his graft if he/she started dialysis and was not able to subsequently be removed from dialysis or underwent graft nephrectomy.
Time Frame: Baseline to end of study (Month 24)
Population: Safety population: All randomized subjects who took at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Upper Everolimus Blood Target + Very Low Dose Cyclosporine | Standard Everolimus Blood Target + Low Dose Cyclosporine
Number analyzed (Participants) | 142 | 143
Participants
  Died | 2 | 3
  Lost graft | 6 | 15
  Died or lost graft | 8 | 18

4. Secondary Outcome: Number of Participants With Adverse Events (AE), Serious Adverse Events (SAE) or Deaths
Description: Safety was assessed using reports of adverse events of all participants in this study. Serious adverse events are those events that resulted in death, were life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or was a congenital anomaly/birth defect.
Time Frame: Baseline to end of study (Month 24)
Population: Safety population: All randomized subjects who took at least one dose of study drug.
Measure: Number; unit: Partcipants
Arm/Group | Upper Everolimus Blood Target + Very Low Dose Cyclosporine | Standard Everolimus Blood Target + Low Dose Cyclosporine
Number analyzed (Participants) | 142 | 143
Partcipants
  AEs | 142 | 143
  Infection | 95 | 101
  Clinically significant AEs | 58 | 53
  SAEs | 85 | 90
  Died | 2 | 3

ADVERSE EVENTS:
Time Frame: 24 months
Description: Population includes all the enrolled patients in the overall core and extension study.
Arm/Group | Upper Everolimus Blood Target + Very Low Dose Cyclosporine | Standard Everolimus Blood Target + Low Dose Cyclosporine
Serious Adverse Events (participants affected / at risk) | 85/142 | 90/143
Other Adverse Events (participants affected / at risk) | 142/142 | 142/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Upper Everolimus Blood Target + Very Low Dose Cyclosporine (N=142) | Standard Everolimus Blood Target + Low Dose Cyclosporine (N=143)
Anaemia (Blood and lymphatic system disorders) | 3 | 5
Bone marrow toxicity (Blood and lymphatic system disorders) | 1 | 0
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Cardiovascular disorder (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1
Pulmonary arteriovenous fistula (Congenital, familial and genetic disorders) | 0 | 1
Orbital oedema (Eye disorders) | 0 | 1
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 2
Intestinal perforation (Gastrointestinal disorders) | 0 | 2
Malabsorption (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Implant site effusion (General disorders) | 1 | 0
Inflammation (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 2
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 13 | 17
Sudden death (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 1
Kidney transplant rejection (Immune system disorders) | 11 | 9
Transplant rejection (Immune system disorders) | 7 | 12
Abdominal abscess (Infections and infestations) | 1 | 0
Bronchitis acute (Infections and infestations) | 1 | 1
Bronchopneumonia (Infections and infestations) | 1 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 3 | 3
Ear infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 2
Gastroenteritis bacterial (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Infected lymphocele (Infections and infestations) | 1 | 1
Omphalitis (Infections and infestations) | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 4
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 2 | 1
Relapsing fever (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 7 | 4
Urosepsis (Infections and infestations) | 2 | 0
Viral infection (Infections and infestations) | 0 | 2
Wound infection (Infections and infestations) | 1 | 0
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0
Chronic allograft nephropathy (Injury, poisoning and procedural complications) | 3 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 0 | 5
Drug toxicity (Injury, poisoning and procedural complications) | 2 | 1
Graft dysfunction (Injury, poisoning and procedural complications) | 0 | 2
Injury (Injury, poisoning and procedural complications) | 1 | 0
Kidney rupture (Injury, poisoning and procedural complications) | 2 | 1
Perinephric collection (Injury, poisoning and procedural complications) | 1 | 0
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 | 2
Arterial bruit (Investigations) | 1 | 0
Biopsy endometrium (Investigations) | 0 | 1
Blood creatine increased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 13 | 7
Blood culture positive (Investigations) | 1 | 0
Blood pressure decreased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 0 | 1
Creatine urine increased (Investigations) | 1 | 0
Cytomegalovirus test (Investigations) | 0 | 1
Legionella serology (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Epithelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 1 | 0
Anuria (Renal and urinary disorders) | 2 | 1
Calculus bladder (Renal and urinary disorders) | 0 | 1
Diffuse mesangial sclerosis (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Focal glomerulosclerosis (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 2 | 2
Hydronephrosis (Renal and urinary disorders) | 1 | 2
Nephritis interstitial (Renal and urinary disorders) | 1 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 1 | 2
Proteinuria (Renal and urinary disorders) | 2 | 2
Renal artery stenosis (Renal and urinary disorders) | 1 | 4
Renal failure acute (Renal and urinary disorders) | 4 | 1
Renal impairment (Renal and urinary disorders) | 3 | 6
Renal tubular necrosis (Renal and urinary disorders) | 1 | 1
Ureteral disorder (Renal and urinary disorders) | 0 | 1
Ureteric stenosis (Renal and urinary disorders) | 2 | 3
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 1
Urogenital fistula (Renal and urinary disorders) | 1 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 2 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 2
Ovarian cyst torsion (Reproductive system and breast disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cholecystectomy (Surgical and medical procedures) | 0 | 1
Inguinal hernia repair (Surgical and medical procedures) | 1 | 0
Lymphocele marsupialisation (Surgical and medical procedures) | 0 | 1
Nephrectomy (Surgical and medical procedures) | 0 | 1
Nephrostomy (Surgical and medical procedures) | 0 | 1
Parathyroidectomy (Surgical and medical procedures) | 1 | 0
Removal of ambulatory peritoneal catheter (Surgical and medical procedures) | 0 | 1
Stent removal (Surgical and medical procedures) | 0 | 1
Ureteric repair (Surgical and medical procedures) | 0 | 1
Aneurysm (Vascular disorders) | 0 | 4
Arteriovenous fistula (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 4 | 3
Haemorrhage (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 2 | 2
Hypotension (Vascular disorders) | 1 | 1
Lymphocele (Vascular disorders) | 12 | 5
Lymphorrhoea (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Upper Everolimus Blood Target + Very Low Dose Cyclosporine (N=142) | Standard Everolimus Blood Target + Low Dose Cyclosporine (N=143)
Anaemia (Blood and lymphatic system disorders) | 82 | 73
Leukopenia (Blood and lymphatic system disorders) | 13 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 7
Tachycardia (Cardiac disorders) | 9 | 3
Constipation (Gastrointestinal disorders) | 18 | 11
Diarrhoea (Gastrointestinal disorders) | 18 | 18
Oedema peripheral (General disorders) | 37 | 36
Pyrexia (General disorders) | 32 | 40
Kidney transplant rejection (Immune system disorders) | 3 | 10
Cytomegalovirus infection (Infections and infestations) | 5 | 13
Urinary tract infection (Infections and infestations) | 69 | 81
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 23 | 31
Blood creatinine increased (Investigations) | 17 | 12
Transaminases increased (Investigations) | 12 | 9
Weight increased (Investigations) | 9 | 9
Acidosis (Metabolism and nutrition disorders) | 11 | 7
Diabetes mellitus (Metabolism and nutrition disorders) | 12 | 7
Dyslipidaemia (Metabolism and nutrition disorders) | 66 | 55
Fluid retention (Metabolism and nutrition disorders) | 13 | 8
Hypercholesterolaemia (Metabolism and nutrition disorders) | 23 | 24
Hyperglycaemia (Metabolism and nutrition disorders) | 15 | 11
Hyperkalaemia (Metabolism and nutrition disorders) | 7 | 9
Hyperlipidaemia (Metabolism and nutrition disorders) | 27 | 26
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 21 | 17
Hyperuricaemia (Metabolism and nutrition disorders) | 30 | 30
Hypocalcaemia (Metabolism and nutrition disorders) | 33 | 19
Hypokalaemia (Metabolism and nutrition disorders) | 23 | 31
Iron deficiency (Metabolism and nutrition disorders) | 2 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 4
Anxiety (Psychiatric disorders) | 5 | 8
Proteinuria (Renal and urinary disorders) | 18 | 12
Renal tubular necrosis (Renal and urinary disorders) | 12 | 10
Ovarian cyst (Reproductive system and breast disorders) | 9 | 4
Hypertension (Vascular disorders) | 32 | 29
Lymphocele (Vascular disorders) | 21 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.